CLINICAL TRIAL: NCT01487629
Title: Bevacizumab Versus Ranibizumab for Refractory Diabetic Macular Edema
Brief Title: Bevacizumab Versus Ranibizumab for the Treatment of Diabetic Macular Edema
Acronym: IBERA-DME
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Rodrigo Jorge, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13368/2010
Record Dates: First submitted 2011-12-02; First posted 2011-12-07 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Diabetic Retinopathy; Macular Edema
Keywords: Diabetic Retinopathy; Macular Edema; Bevacizumab; Ranibizumab
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema | interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bevacizumab (Experimental): Treatment of macular edema with intravitreal Bevacizumab
  Interventions: Drug: Bevacizumab
- Ranibizumab (Experimental): Treatment of macular edema with intravitreal Ranibizumab
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab, 1.5 mg, intravitreal, throughout the study
  Other Names: Avastin
  Arms: Bevacizumab
Drug: Ranibizumab — Ranibizumab, 0.5 mg, intravitreal, throughout the study
  Other Names: Lucentis
  Arms: Ranibizumab

SUMMARY:
The purpose of this study is to compare the morphological and visual acuity outcomes associated with 1.5 mg bevacizumab versus 0.5 ranibizumab intravitreal injections for treatment of diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Center-involving Diabetic macular edema unresponsive to LASER therapy performed at least 3 moths prior to inclusion;
* Best corrected visual acuity equal or worse than 20/40 and better than 20/800;
* Central subfield macular thickness greater than 300 µm

Exclusion Criteria:

* Aphakia
* High-risk proliferative diabetic retinopathy
* Previous treatment for DME in the past three months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-04; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Central subfield macular thickness (CSFT) change | Monthly from baseline to Week 48
  Central subfield macular thickness (CSFT) measured with spectral-domain optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Best-corrected visual acuity change | Monthly from baseline to week 48
  Best-corrected visual acuity using ETDRS charts

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Jorge, MD, PhD, Principal Investigator — University of Sao Paulo; Felipe Almeida, MD, Study Director — Hospital das Clinicas - Faculdade de Medicina de Ribeirão Preto
Locations (1):
- Clinics Hospital of Ribeirão Preto, School of Medicine of Ribeirão Preto, USP, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Nepomuceno AB, Takaki E, Paes de Almeida FP, Peroni R, Cardillo JA, Siqueira RC, Scott IU, Messias A, Jorge R. A prospective randomized trial of intravitreal bevacizumab versus ranibizumab for the management of diabetic macular edema. Am J Ophthalmol. 2013 Sep;156(3):502-510.e2. doi: 10.1016/j.ajo.2013.04.026. Epub 2013 Jun 21. PMID 23795985